CLINICAL TRIAL: NCT02145182
Title: A Randomized, Parallel-group, Double-blind, Placebo-controlled, Multi-center Study of Eculizumab for the Prevention of Delayed Graft Function After Kidney Transplantation in Adult Subjects at Increased Risk of Delayed Graft Function.
Brief Title: Prevention of Delayed Graft Function Using Eculizumab Therapy (PROTECT Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ECU-DGF-201; 2013-004650-25 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-05-22 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Delayed Graft Function
Keywords: DGF; Dialysis; Kidney; Kidney Transplantation; eGFR; Complement; Eculizumab
MeSH Terms: conditions — Delayed Graft Function | interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Eculizumab was administered by intravenous (IV) infusion over 25-45 minutes (min) for 2 doses (on the day of transplant then 18-24 hours [h] later).
  Interventions: Drug: Eculizumab
- Placebo (Placebo Comparator): Placebo was administered by IV infusion over 25-45 min for 2 doses (on the day of transplant then 18-24 h later).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eculizumab — Eculizumab is a complement component 5 inhibitor.
  Other Names: Soliris
  Arms: Active
Drug: Placebo — 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine if eculizumab is safe and could be used to prevent delayed graft function (DGF) following kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* Has dialysis-dependent renal failure (initiated more than 2 months prior to transplant)
* Participant is to receive a first kidney transplant from a standard criteria donor or expanded criteria donor deceased donor with a DGF risk score using the Irish scale of ≥25% (to be determined prior to surgery and before randomization)
* Able to provide written informed consent
* Willing and able to comply with the requirements of the study protocol
* Female participants of child-bearing potential must have a negative serum pregnancy test (serum beta-human chorionic gonadotropin) and must be practicing an effective, reliable, and medically approved contraceptive regimen at the time of consent and for up to 5 months following discontinuation of treatment

Exclusion Criteria:

* Participant to receive a multi-organ transplant
* Participant to receive kidney(s) from donors <6 years of age
* Participant to receive a dual kidney transplant (from same donor, including en bloc)
* Participant to receive a living donor kidney
* Participant is highly sensitized (high risk to develop acute antibody-mediated rejection) to the donor (as determined by local center practice). Testing to determine high risk may include but is not limited to flow cytometric cross match, single antigen bead testing and/or complement dependent cytotoxicity
* Participant has received a previous transplant
* Participant is participating in another investigational study
* Participant has a body mass index >40 kilograms/square meter at screening
* Participant will be the recipient of an A, B, O Blood Glycoproteins (ABO) (blood type) incompatible kidney (A2 donors to B and O recipients will be allowed if the site has the ability to confirm A2 subtype)
* Participant will receive a kidney from a donation after cardiac death donor
* Participant has a predicted Irish model risk of DGF <25%
* Female participants who are pregnant or breast feeding
* Female participants of child bearing potential who are unable or unwilling to use a medically acceptable form of contraception
* Participants with a history of human immunodeficiency virus, or active hepatitis C virus or hepatitis B virus infection
* Participants with active bacterial or other infection which is clinically significant in the opinion of the Investigator
* Participants with a history of splenectomy
* Participants with unresolved meningococcal disease
* Participants with an unresolved systemic bacterial or fungal infection
* Participants with known or suspected hereditary complement deficiency (for example, but not limited to: atypical hemolytic uremic syndrome, paroxysmal nocturnal hemoglobinuria)
* Participant has a current malignancy or a history of any malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix that has been treated appropriately
* Participant has a history of or is believed by the Investigator to have used an illicit drug(s) and/or abused alcohol within 3 months prior to screening
* Participant has a psychiatric or physical illness that in the opinion of the Investigator would interfere with the ability of the participant to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2014-08-21 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (30):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - Palo Alto, California
  - San Francisco, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Livingston, New Jersey
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Charleston, South Carolina
  - Fort Worth, Texas
  - Houston, Texas
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Australia (4):
  - Camperdown, New South Wales
  - Westmead, New South Wales
  - Adelaide, South Australia
  - Clayton, Victoria
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil
- Canada (4):
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec
- Prague, Czechia
- France (10):
  - Bordeaux
  - Créteil
  - Le Kremlin-Bicêtre
  - Lyon
  - Nantes
  - Paris
  - Strasbourg
  - Suresnes
  - Toulouse
  - Tours
- Germany (8):
  - Berlin
  - Dresden
  - Erlangen
  - Essen
  - Hamburg
  - Hannoversch Münden
  - Hanover
  - Kiel
- Italy (6):
  - Bari
  - Brescia
  - Milan
  - Padua
  - Torino
  - Verona
- Spain (7):
  - Badalona
  - Barcelona
  - Madrid
  - Santander
  - Seville
  - Valencia
  - Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-nine centers in Australia, Brazil, Canada, Czech Republic, France, Germany, Italy, Spain, and the United States of America participated in this study. The study recruited participants who had been receiving dialysis for a median of approximately 50 months before undergoing transplantation and received a kidney from a deceased donor.
Pre-assignment Details: Written consent was provided prior to study-required assessments (N=333). Participants who passed screening (N=314) were vaccinated against Neisseria meningitidis. A total of 314 were randomized; of these, 286 underwent transplantation and received eculizumab or placebo. Two participants received placebo but withdrew prior to transplantation.
Groups:
- Eculizumab: Participants received 2 doses of eculizumab: the first dose was just prior to reperfusion of the allograft and the second dose was within 18 to 24 hours (h) of completion of administration of the first dose. Each dose of eculizumab was administered by intravenous (IV) infusion over 25 to 45 minutes (min). The first dose was 1200 milligrams (mg) in 240 milliliters (mL) (5 mg/mL); the second dose was 900 mg in 180 mL (5 mg/mL).
- Placebo: Participants received 2 doses of placebo (0.9% sodium chloride [NaCl]): the first dose was just prior to reperfusion of the allograft and the second dose was within 18 to 24 h of completion of administration of the first dose. Each dose of placebo was administered by IV infusion over 25 to 45 min. The first dose was 240 mL of 0.9% NaCl; the second dose was 180 mL of 0.9% NaCl.
Period: Overall Study
Arm/Group | Eculizumab | Placebo
Started | 142 | 146
Received at Least 1 Dose of Study Drug | 142 | 146
Completed | 124 | 130
Not Completed | 18 | 16
Not completed — Adverse Event | 4 | 1
Not completed — Death | 7 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Pre-transplant Withdrawal | 0 | 2
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Population: Safety Set: all participants who received at least 1 dose of study drug (placebo or eculizumab).
Groups:
- Eculizumab: Participants received 2 doses of eculizumab: the first dose was just prior to reperfusion of the allograft and the second dose was within 18 to 24 h after completion of administration of the first dose. Eculizumab was administered by IV infusion over 25 to 45 min for each dose. The first dose was 1200 mg in 240 mL (5 mg/mL); the second dose was 900 mg in 180 mL (5 mg/mL).
- Placebo: Participants received 2 doses of placebo: the first dose was just prior to reperfusion of the allograft and the second dose was within 18 to 24 h after completion of administration of the first dose. Placebo was administered by IV infusion over 25 to 45 min for each dose. The first dose was 240 mL of 0.9% NaCl; the second dose was 180 mL of 0.9% NaCl.
- Total: Total of all reporting groups
Arm/Group | Eculizumab | Placebo | Total
Number analyzed (Participants) | 142 | 146 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.29) | 57.1 (13.03) | 57.3 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 92
  Male | 95 | 101 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 23 | 46
  Not Hispanic or Latino | 108 | 113 | 221
  Unknown or Not Reported | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 2 | 3
  Asian | 0 | 4 | 4
  Black or African American | 38 | 37 | 75
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 88 | 92 | 180
  Other | 9 | 7 | 16
  Multiple | 1 | 1 | 2
  Unknown | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants With Delayed Graft Function (DGF) In The First Seven Days Post-transplant
Description: Results are reported for the DGF composite endpoint, defined as the occurrence of DGF (dialysis for any reason in the first 7 days post transplantation), graft loss, death, or loss to follow-up (including discontinuation) in the first 7 days post transplantation and for each item of the composite endpoint. Loss to follow-up included withdrawal due to any reason other than death. The sum of the counts in the events that make up the DGF composite may be greater than the composite count, because a participant who experienced multiple events was only counted once in the composite.
Time Frame: First 7 days post transplantation
Population: Full Analysis Set: all participants who were randomized to treatment and received a deceased donor kidney transplant and at least 1 dose of study drug (placebo or eculizumab).
Measure: Number; unit: percentage of participants
Groups:
- Eculizumab: Participants received 2 doses of eculizumab: the first dose was just prior to reperfusion of the allograft and the second dose was within 18 to 24 h of completion of administration of the first dose. Each dose of eculizumab was administered by IV infusion over 25 to 45 min. The first dose was 1200 mg in 240 mL (5 mg/mL); the second dose was 900 mg in 180 mL (5 mg/mL).
- Placebo: Participants received 2 doses of placebo: the first dose was just prior to reperfusion of the allograft and the second dose was within 18 to 24 h of completion of administration of the first dose. Each dose of placebo was administered by IV infusion over 25 to 45 min. The first dose was 240 mL of 0.9% NaCl; the second dose was 180 mL of 0.9% NaCl.
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 142 | 144
percentage of participants
  DGF Composite | 35.9 | 41.7
  DGF | 33.8 | 39.6
  Death | 0.0 | 1.4
  Graft Loss | 0.7 | 3.5
  Lost to Follow-up (including discontinuation) | 3.5 | 1.4
Statistical Analysis 1: Comparison: Eculizumab vs Placebo; Analysis of DGF composite; Test type: Superiority; p = 0.3983, Regression, Logistic; Logistic regression results for the DGF composite, the effect of treatment adjusted for preservation type, donor type, and Irish score; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.49 to 1.33] — Calculated using the logistic regression model

2. Secondary Outcome: Percentage Of Participants With DGF, Functional DGF, And Immediate Graft Function
Description: DGF was defined as a requirement for dialysis for any reason in the first 7 days post transplantation; functional DGF was defined as no need for dialysis during the first 7 days post transplantation and either (1) a <70% reduction in serum creatinine during the first 7 days post transplantation, or (2) failure of serum creatinine to decrease by at least 10% daily on 3 consecutive days, both measured during the first 7 days post transplantation. Blood and urine samples were collected, but because the study failed to demonstrate a treatment effect and the program subsequently lost funding, the collected data from the samples could not be analyzed to generate summary level data. As such, the data set for this secondary outcome measure cannot be summarized.
Time Frame: First 7 days post transplantation
Population: Full Analysis Set: all participants who were randomized to treatment and received a deceased donor kidney transplant and at least 1 dose of study drug (placebo or eculizumab). Because the study failed to demonstrate a treatment effect and the program subsequently lost funding, collected data could not be analyzed to generate summary level data.
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage Of Participants Who Required Dialysis Post Transplantation
Description: The need for dialysis was assessed by evaluation of renal function; this included urine volume, blood urea nitrogen, serum creatinine, and, starting on Day 2, the creatinine reduction ratio. Blood and urine samples were collected, but because the study failed to demonstrate a treatment effect and the program subsequently lost funding, the collected data from the samples could not be analyzed to generate summary level data. As such, the data set for this secondary outcome measure cannot be summarized.
Time Frame: First 30 days post transplantation
Population: as for outcome 2
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: The eGFR was calculated by using the Modification of Diet in Renal Disease 7 equation at Day 28 post transplantation. The equation requires serum creatinine, age, ethnicity, gender, blood urea nitrogen, and albumin. The eGFR was calculated retrospectively from participant demographics and laboratory chemistries and is reported in mL/min/square meter (m^2).
Time Frame: Day 28 post transplantation
Population: Safety Set: all participants who received at least 1 dose of study drug (placebo or eculizumab) and made the Day 28 visit.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 132 | 135
mL/min/1.73 m^2 | 42.640 (20.7491) | 39.954 (20.3288)

5. Secondary Outcome: Percentage Of Participants With Rejection-free Graft Survival
Description: Graft survival was defined as not having biopsy-proven acute rejection per Banff criteria, graft loss, or participant death. Participants who did not experience graft loss or death were censored at 365 days or the day they withdrew, whichever came first. There were no time-specific protocol mandated biopsies. Kidney biopsy would have been performed for cause at the discretion of the Investigator to assess poor graft function and would have been obtained prior to initiating treatment of suspected allograft rejection. Only summaries of Kaplan-Meier estimates of graft survival at Week 26 (Month 6) and Week 52 (Month 12) are reported.
Time Frame: Week 26 and 52 post transplantation
Population: Full Analysis Set: all participants who were randomized to treatment and received a deceased donor kidney transplant and at least 1 dose of study drug (placebo or eculizumab). Eculizumab participants censored: Month 6 = 7; Month 12 = 132. Placebo participants censored: Month 6 = 2; Month 12 = 128.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eculizumab | Placebo
Number analyzed (Participants) | 142 | 144
percentage of participants
  Graft Survival at Month 6 | 94.89 [89.58 to 97.53] | 90.96 [84.94 to 94.65]
  Graft Survival at Month 12 | 92.66 [86.78 to 95.98] | 88.69 [82.17 to 92.92]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were required to be reported during the study up to 60 days after the last dose of study drug and serious adverse events were required to be reported during the study through 12 months of follow-up.
Arm/Group | Eculizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 8/142 | 7/146
Serious Adverse Events (participants affected / at risk) | 92/142 | 102/146
Other Adverse Events (participants affected / at risk) | 139/142 | 142/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=142) | Placebo (N=146)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 3
Angina unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Internal hernia (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 1
Pyrexia (General disorders) | 4 | 4
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0
Kidney transplant rejection (Immune system disorders) | 4 | 3
Renal transplant failure (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 2 | 0
Bronchitis moraxella (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 3 | 2
Cytomegalovirus viraemia (Infections and infestations) | 3 | 3
Diabetic foot infection (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 3
Enterococcal infection (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 3 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 3 | 0
Gangrene (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 2 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 8
Pneumonia cytomegaloviral (Infections and infestations) | 2 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 2 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 4
Respiratory tract infection (Infections and infestations) | 2 | 1
Salmonella sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 4 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 4
Urinary tract infection bacterial (Infections and infestations) | 3 | 2
Urinary tract infection enterococcal (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 6 | 3
Wound abscess (Infections and infestations) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 4 | 4
Delayed graft function (Injury, poisoning and procedural complications) | 0 | 1
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Graft loss (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Perinephric collection (Injury, poisoning and procedural complications) | 0 | 2
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 3
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Wound decomposition (Injury, poisoning and procedural complications) | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Biopsy kidney abnormal (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 2
Donor specific antibody present (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Neuromyopathy (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 6
Anuria (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 2 | 0
Obstructive nephropathy (Renal and urinary disorders) | 1 | 1
Renal artery dissection (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 3
Renal cyst haemorrhage (Renal and urinary disorders) | 1 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 2 | 3
Renal tubular necrosis (Renal and urinary disorders) | 1 | 2
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 2 | 0
Ureteric stenosis (Renal and urinary disorders) | 2 | 2
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary fistula (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 7
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 3
Lymphocele (Vascular disorders) | 2 | 1
Lymphorrhoea (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 0
Shock (Vascular disorders) | 0 | 2
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=142) | Placebo (N=146)
Anaemia (Blood and lymphatic system disorders) | 77 | 75
Leukocytosis (Blood and lymphatic system disorders) | 8 | 7
Leukopenia (Blood and lymphatic system disorders) | 37 | 30
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 15
Atrial fibrillation (Cardiac disorders) | 9 | 10
Tachycardia (Cardiac disorders) | 17 | 12
Abdominal pain (Gastrointestinal disorders) | 13 | 14
Constipation (Gastrointestinal disorders) | 40 | 40
Diarrhoea (Gastrointestinal disorders) | 37 | 35
Dyspepsia (Gastrointestinal disorders) | 9 | 8
Nausea (Gastrointestinal disorders) | 36 | 32
Vomiting (Gastrointestinal disorders) | 30 | 24
Asthenia (General disorders) | 12 | 20
Chest pain (General disorders) | 6 | 11
Oedema (General disorders) | 7 | 8
Oedema peripheral (General disorders) | 41 | 57
Pyrexia (General disorders) | 26 | 20
Kidney transplant rejection (Immune system disorders) | 14 | 7
BK virus infection (Infections and infestations) | 18 | 18
Cytomegalovirus infection (Infections and infestations) | 17 | 17
Upper respiratory tract infection (Infections and infestations) | 4 | 10
Urinary tract infection (Infections and infestations) | 22 | 33
Procedural pain (Injury, poisoning and procedural complications) | 30 | 21
Blood creatinine increased (Investigations) | 14 | 21
Urine output decreased (Investigations) | 5 | 11
Acidosis (Metabolism and nutrition disorders) | 35 | 24
Decreased appetite (Metabolism and nutrition disorders) | 3 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 12 | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 10 | 15
Fluid overload (Metabolism and nutrition disorders) | 12 | 26
Hypercalcaemia (Metabolism and nutrition disorders) | 11 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 23
Hyperkalaemia (Metabolism and nutrition disorders) | 59 | 67
Hyperphosphataemia (Metabolism and nutrition disorders) | 13 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 33 | 23
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 25
Hypomagnesaemia (Metabolism and nutrition disorders) | 40 | 28
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 28 | 19
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 15
Dizziness (Nervous system disorders) | 5 | 10
Headache (Nervous system disorders) | 13 | 10
Tremor (Nervous system disorders) | 21 | 28
Anxiety (Psychiatric disorders) | 10 | 10
Insomnia (Psychiatric disorders) | 16 | 16
Acute kidney injury (Renal and urinary disorders) | 6 | 10
Bladder spasm (Renal and urinary disorders) | 6 | 8
Dysuria (Renal and urinary disorders) | 14 | 20
Haematuria (Renal and urinary disorders) | 14 | 15
Proteinuria (Renal and urinary disorders) | 8 | 6
Renal tubular necrosis (Renal and urinary disorders) | 15 | 10
Urinary retention (Renal and urinary disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 9
Hypertension (Vascular disorders) | 34 | 39
Hypotension (Vascular disorders) | 29 | 33
Lymphocele (Vascular disorders) | 9 | 4

LIMITATIONS AND CAVEATS:
Because the study failed to demonstrate a treatment effect and the program subsequently lost funding, all collected data could not be analyzed to generate summary level data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No